CLINICAL TRIAL: NCT01147042
Title: Assessment of the Biochemical Response to Interferon-Gamma in Subjects With Specific Gene Mutation in Chronic Granulomatous Disease
Brief Title: Biochemical Response to Interferon-Gamma in Subjects With Specific Gene Mutation in Chronic Granulomatous Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Early termination due to only 2 subjects completing trial.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 100123; 10-I-0123 (Other: National Institutes of Health)
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Results first posted 2017-09-20 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-08

CONDITIONS: IFN-Gamma Therapy; CGD Gene Mutation; CGD Response to IFNg; CGD - Chronic Granulomatous Disease; Immunodeficiency Disease
Keywords: NADPH Oxidase-Nicotinamide Adenine Dinucleotide Phosphate; Chronic Granulomatous Disease; Gene Mutation; Superoxide by Phagocytes; Interferon-Gamma
MeSH Terms: conditions — Granulomatous Disease, Chronic; Immunologic Deficiency Syndromes | interventions — Interferon-gamma

STUDY DESIGN:
Intervention Model Description: Dose frequency increased from once per week to three times per week, the recommended dose frequency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- gp91 CGD with relatively high baseline superoxide (Active Comparator): Patients with X-linked Chronic Granulomatous Disease (CGD) with a missense gp91phox mutation and relatively high baseline superoxide production.
  IFN-gamma was the administered intervention.
  Interventions: Drug: IFN-gamma
- Autosomal Recessive CGD with p47 (Active Comparator): Patients with Autosomal Recessive Chronic Granulomatous Disease (CGD) with p47 phox mutation. IFN-gamma was the administered intervention.
  Interventions: Drug: IFN-gamma

INTERVENTIONS:
Drug: IFN-gamma — Following a washout period subjects have a subcutaneous injection of 50 mcg per meter squared once per week, Monday, for 4 weeks, twice per week, Monday and Thursday, for 4 weeks, then thrice per week, Monday, Wednesday, Friday, for 4 weeks. Total treatment period is 12 weeks.
  Other Names: Interferon-gamma

SUMMARY:
Background:

- Chronic granulomatous disease (CGD) is an immunodeficiency disease in which white blood cells are unable to kill certain bacteria and fungi. People with CGD are more likely to develop recurrent life-threatening infections. Certain changes or mutations in genes contribute to the severity of CGD, and also appear to affect the success of treatment with interferon-gamma, a substance that is used to improve the immune system s ability to fight infection. Researchers are interested in studying changes in the immune system caused by interferon-gamma treatment of CGD in individuals with different mutations that cause CGD.

Objectives:

- To compare changes in the immune system caused by interferon-gamma treatment for CGD in individuals with different mutations that cause CGD.

Eligibility:

- Individuals of any age who have been diagnosed with CGD and have specific types of mutations that cause CGD (to be determined after testing).

Design:

* Participants will be screened with a medical history, physical examination, and blood and urine tests. Participants must weigh more than 11 kilograms (~24 pounds) to participate in the study.
* Participants will receive injections of interferon-gamma once weekly for 4 weeks, twice weekly for 4 weeks, and then three times weekly for 4 weeks (a total of 24 injections).
* Blood will be drawn periodically during treatment and for 8 weeks after the treatment, for a total of 21 weeks on the study. Participants will regularly provide information on their symptoms and responses to treatment to the study researchers.

DETAILED DESCRIPTION:
Chronic Granulomatous Disease (CGD) is caused by mutations of 1 of the 4 proteins comprising the NADPH oxidase that result in decreased or absent production of superoxide by phagocytes, and predisposes CGD subjects to life-threatening infection. Intensive management with antibiotics and antifungal agents has dramatically increased the life expectancy of subjects with CGD. Interferon-gamma (IFN gamma), which increases superoxide production by neutrophils and enhances their antimicrobial activity, is an FDA approved therapy for CGD and is now the standard of care. However, there is substantial variability in the biochemical and clinical response to IFN gamma treatment. Recently, the specific mutations of the genes responsible for causing CGD in most of the subjects followed at the NIH have been characterized. Because of this, it is now known that the severity of the disease is correlated not only with inheritance pattern, but also with the specific underlying mutation. It is not known, however, if the biochemical response to IFN gamma therapy correlates with the specific mutation as well.

Since treatment with IFN gamma is expensive, requires frequent injections, and in some subjects results in systemic side effects, it would be useful to determine whether the biochemical response and systemic side effects correlate with the underlying mutation GCD.

We hypothesize that subjects with X-linked CGD due to nonsense/frameshift/RNA processing/deletion mutations of the gp91phox component of the NADPH oxidase will generate a smaller biochemical response to IFN gamma therapy compared to subjects with missense gp91phox mutations or the autosomal recessive form of CGD that results from mutations of the p47phox or p67phox components.

The primary objective of this study is to assess the predictability of IFN gamma responsiveness in CGD based on mutational analysis. compare the change in function of the NADPH oxidase during treatment with an escalating dose of IFN gamma in subjects with CGD resulting from missense or nonsense/frameshift/RNA processing/deletion gp91phox mutations or mutations of p47phox or p67phox. The secondary objectives are to assess changes in superoxide production, expression of NADPH oxidase components, neutrophil bactericidal capacity for Staphyloccus aureus, cytokines, cell surface markers, antibodies, lymphocyte subsets, constitutional symptoms , and gene expression in leukocytes from subjects with missense gp91phox mutations, nonsense/frameshift/RNA processing/deletion gp91phox mutations, p47phox mutations, and p67phox mutations after treatment with IFN gamma to assess changes in the expression of NADPH oxidase components, cytokines, cell surface markers, antibody production, production of various lymphocyte subsets, constitutional symptoms and gene expression in leukocytes from these subjects following treatment with IFN gamma. This knowledge will assist physicians in determining which subjects are likely to respond to full dose and alternative dose therapy with IFN gamma and provide information about biochemical responses of to these regimens in subjects with specific CDG gene mutations enabling them to better counsel and manage subjects with CGD.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects may be enrolled if they are:

1. Already are enrolled on an existing CGD protocol at the Clinical Center (and will remain enrolled on their existing protocol);
2. Are included in one of the study cohorts listed below;
3. Male or female;
4. Able to comply with self-administration of a subcutaneous injection; and
5. Willing to have their blood samples stored for the duration of this study and for future research.

Study Groups/Cohorts:

X-linked CGD Nonsense/Frameshift/RNA Processing/Deletion Mutations Cohort: Subjects in this cohort must have X-linked CGD resulting from a documented nonsense, frameshift, RNA processing, or deletion gene mutation. Subjects with other gene defects or for whom the specific genetic defect has not been determined are not eligible for inclusion in this cohort.

X-linked CGD Missense Mutation with Low Baseline Superoxide Production (less than or equal to 2.5 nmol/10(6) cells/hr) Cohort: Subjects in this cohort must have X-linked CGD resulting from a documented missense gene and superoxide production by cytochrome c reduction assay at baseline of less than or equal to 2.5 nmol/10(6) cells/hr. Subjects with other gene defects or for whom the specific genetic defect has not been determined are not eligible for inclusion in this cohort.

X-linked CGD Missense Mutation with Higher Baseline Superoxide Production (greater than 2.5 nmol/10(6) cells/hr) Cohort: Subjects in this cohort must have X-linked CGD resulting from a documented missense gene and superoxide production by cytochrome c reduction assay at baseline of greater than 2.5 nmol/10(6) cells/hr. Subjects with other gene defects or for whom the specific genetic defect has not been determined are not eligible for inclusion in this cohort.

Autosomal Recessive p47phox CGD Cohort: Subjects in this cohort must have autosomal recessive CGD resulting from a documented p47phox gene mutation. Subjects with other gene defects or for whom the specific genetic defect has not been determined are not eligible for inclusion in this cohort.

Autosomal Recessive p67phox CGD Cohort: Subjects in this cohort must have autosomal recessive CGD resulting from a documented p67phox gene mutation. Subjects with other gene defects or for whom the specific genetic defect has not been determined are not eligible for inclusion in this cohort.

EXCLUSION CRITERIA:

Subjects are excluded from the study who:

1. Have undergone successful bone marrow transplantation;
2. Had a serious adverse reaction to IFN gamma in the past;
3. Are pregnant or breast feeding;
4. Weigh less than 11 kg;
5. Are currently on therapy with INF gamma;
6. Have any of the following medical conditions:

   * Coronary artery disease;
   * Hepatic disease and/or liver enzymes elevated above 3 times normal;
   * Seizure disorder, or
   * Severe myelosuppression (absolute neutrophil count less than1000 cells/mm(3)).

Participation of Minors: minor patients will be invited to participant in this study.

Participation of Women: Exposure to IFN gamma by the developing human fetus may be detrimental. For this reason, women of childbearing-age will have a pregnancy test prior to undergoing study procedures. Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should immediately inform study staff and her primary care physician.

Pregnancy and Lactation: The effects of IFN gamma therapy on the developing fetus and newborn infant have not been studied. Therefore, it is not recommended that subjects who are pregnant or breast-feeding receive IFN gamma and they will be excluded from this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-05-18; Primary Completion 2014-11-14 (Actual); Study Completion 2014-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John I Gallin, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Winkelstein JA, Marino MC, Johnston RB Jr, Boyle J, Curnutte J, Gallin JI, Malech HL, Holland SM, Ochs H, Quie P, Buckley RH, Foster CB, Chanock SJ, Dickler H. Chronic granulomatous disease. Report on a national registry of 368 patients. Medicine (Baltimore). 2000 May;79(3):155-69. doi: 10.1097/00005792-200005000-00003. PMID 10844935
- [Background] Nathan CF, Murray HW, Wiebe ME, Rubin BY. Identification of interferon-gamma as the lymphokine that activates human macrophage oxidative metabolism and antimicrobial activity. J Exp Med. 1983 Sep 1;158(3):670-89. doi: 10.1084/jem.158.3.670. PMID 6411853
- [Background] Berton G, Zeni L, Cassatella MA, Rossi F. Gamma interferon is able to enhance the oxidative metabolism of human neutrophils. Biochem Biophys Res Commun. 1986 Aug 14;138(3):1276-82. doi: 10.1016/s0006-291x(86)80421-1. PMID 3092821
- [Background] International Chronic Granulomatous Disease Cooperative Study Group. A controlled trial of interferon gamma to prevent infection in chronic granulomatous disease. N Engl J Med. 1991 Feb 21;324(8):509-16. doi: 10.1056/NEJM199102213240801. PMID 1846940

RESULTS

PARTICIPANT FLOW:
Groups:
- gp91 CGD With HIGH Baseline Superoxide: Patients with X-linked Chronic Granulomatous Disease (CGD) with a missense gp91phox mutation and relatively high baseline superoxide production
- Autosomal Recessive CGD With p47: Patients with Autosomal Recessive Chronic Granulomatous Disease (CGD) with p47 phox mutation
Period: Overall Study
Arm/Group | gp91 CGD With HIGH Baseline Superoxide | Autosomal Recessive CGD With p47
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- gp91 CGD With Relatively High Baseline Superoxide: Subjects in this cohort have X-linked CGD resulting from a documented missense gene and superoxide production by cytochrome c reduction assay at baseline of greater than 2.5 nmol/106 cells per hour.
  Following a washout period subjects have a subcutaneous injection of 50 mcg per meter squared administered once per week, Monday, for 4 weeks, twice per week, Monday and Thursday, for 4 weeks, then thrice per week, Monday, Wednesday, Friday, for 4 weeks for a total of 12 weeks of Interferon-gamma treatment.
- Autosomal Recessive CGD With p47: Subjects in this cohort have autosomal recessive CGD resulting from a documented p47phox gene mutation.
  Subjects will then be started on a 12 week course of IFN treatment. Subjects will have a subcutaneous injection of 50 mcg/m2 once per week (Monday) for 4 weeks, twice per week (Monday and Thursday) for 4 weeks, then thrice per week (Monday, Wednesday, Friday) for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | gp91 CGD With Relatively High Baseline Superoxide | Autosomal Recessive CGD With p47 | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Basal and PMA-stimulated O2 Production Detected by Ferricytochrome c Reduction in Neutrophils
Time Frame: 21 weeks
Population: Data were not collected.
Arm/Group | gp91 CGD With HIGH Baseline Superoxide | Autosomal Recessive CGD With p47
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- gp91 CGD With Relatively High Baseline Superoxide: Patients with X-linked Chronic Granulomatous Disease (CGD) with a missense gp91phox mutation and relatively high baseline superoxide production
Arm/Group | gp91 CGD With Relatively High Baseline Superoxide
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Early termination due to only 2 subjects completing trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes